CLINICAL TRIAL: NCT01214551
Title: Exercise-induced Bronchoconstriction Diagnostics: Impact of a Repeated Exercise Challenge Test
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Klinikk for allergi og luftveissykdommer (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2010/1551-4
Record Dates: First submitted 2010-09-23; First posted 2010-10-05 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Exercise Induced Bronchoconstriction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to increase the knowledge of the possible diagnostic effect of exercise induced bronchoconstriction performing a repeated exercise challenge test.

DETAILED DESCRIPTION:
Prior studies have shown that the intensity influences the sensitivity of exercise challenge tests (ECT) and that a heart rate-based protocol does not ensure sufficient exercise intensity to induce bronchoconstriction. It is not common clinical practice to perform a pre ECT to establish maximal heart rate or maximal oxygen uptake. The heart rate formula recommended by ATS (HRmax= 220-age) is usually applied to determine recommended intensity of the ECT. Conducting a second ECT, based on the knowledge of the first test, introduce the possibility to adjust the intensity on an individual basis. In addition, based on clinical experience, patients may seem reluctant to perform maximal the first time they undergo an ECT on a treadmill. The hypothesis is that patients are less reluctant to perform maximal the second time they undergo the test when they are more accustomed to the procedure and the treadmill by itself.

ELIGIBILITY:
Inclusion Criteria:

* Referred to Klinikk for allergi og luftveissykdommer
* Meet at least 3 out of 5 criteria (symptoms related to exercise):

  1. Cough during exercise or within 5 minutes after exercise
  2. Wheeze during exercise or within 5 minutes after exercise
  3. Heavy breathing, expiratory in particular, during exercise or within 5 minutes after exercise (duration 5 minutes or more)
  4. Improvement of physical fitness/breath is lacking despite of exercise intensification
  5. Chest tightness during or after exercise
* Patients former diagnosed with-and treated for asthma who have symptoms of EIB are included in the study.

Exclusion Criteria:

* Ongoing respiratory infection or recent respiratory infection, judged by the responsible doctor to be of importance of the result
* The inability to perform an Exercise challenge test with maximum effort

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects referred to Klinikk for allergi og luftveissykdommer
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | up to 4 weeks

SECONDARY OUTCOMES:
Forced vital capacity (FVC) | up to 4 weeks
Forced expiratory flow at 50 % FVC(FEF50%) | up to 4 weeks
Fractional exhaled nitric oxide (FENO) | up to 4 weeks
Total lung capacity (TLC) | up to 4 weeks
Specific airway resistance (sRAW) | up to 4 weeks
Specific airway conductance (sGAW) | up to 4 weeks
Residual volume (RV) | up to 4 weeks
Diffusing capacity (TLCO) | up to 4 weeks
Maximum voluntary ventilation (MVV) | up to 4 weeks
Breathing reserve (BR) | up to 4 weeks
Respiratory exchange ration (RER) | up to 4 weeks
Oxygen uptake peak (VO2 peak) | up to 4 weeks
Heart rate peak (HR peak) | up to 4 weeks
Ventilation peak (VE peak) | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liv B Augestad, Professor, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Klinikk for allergi og luftveissykdommer, Oslo, Ullevål, Norway

REFERENCES:
- [Result] Angell MR, Augestad LB, Haugen TS, Frostad A, Grønnerød TA, Stensrud T. Exercise-induced bronchoconstriction diagnostics: Impact of a repeated exercise challenge test. Open Journal of Respiratory Diseases 4:55-63, 2014 http://file.scirp.org/pdf/OJRD_2014043017202072.pdf